CLINICAL TRIAL: NCT01040663
Title: Isocaloric Dietary Interventions for Insulin Resistance and the Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LNE-0673
Record Dates: First submitted 2009-12-24; First posted 2009-12-29 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dash Diet (Other): Subjects receive DASH diet for 4 weeks
  Interventions: Other: Dietary intervention
- Low GI Diet (Other): Subjects will receive Low GI diet for 4 weeks
  Interventions: Other: Dietary intervention
- Western Style Diet (Other): Subjects will receive western style diet for 4 weeks
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — Subjects will be randomly assigned to receive 1 of 3 diets for 4 weeks.

SUMMARY:
In recent decades, the prevalence of obesity has increased dramatically in the United States. Obesity has been associated with an increased risk of the metabolic syndrome, which is characterized by a cluster of metabolic derangements, including insulin resistance, high blood sugar, high triglycerides, low high density lipoprotein (HDL) cholesterol levels, high blood pressure, and inflammation. Lifestyle interventions, including dietary modification, physical activity, and weight loss, form the basis of treatment for individuals with the metabolic syndrome. However, the optimal composition of the diet is not known at this time. Furthermore, due to hormonal and metabolic changes that accompany weight loss, most people find it very difficult to maintain significant weight reductions over time. As a result, weight regain is exceedingly common.

DETAILED DESCRIPTION:
Several dietary patterns, including the Dietary Approaches to Stop Hypertension study diet (the DASH diet) and the low glycemic index diet (low GI diet), may be useful in the treatment of individuals with the metabolic syndrome, even if body weight stays the same. Novel findings from our own pilot study suggest that these dietary patterns may improve insulin resistance and some other features of the metabolic syndrome, even after just two weeks and in the absence of weight loss. In this important follow-up study, the metabolic effects of the DASH diet and the low GI diet will be compared to those of an Western-style control diet. At least 39 overweight, insulin-resistant volunteers with the metabolic syndrome will be studied during a 32-day inpatient admission. All food will be provided, and body weight will be kept stable throughout the study. Subjects will first undergo testing after consuming a Western-style diet for two weeks. They will then be randomized to one of three study diets: the DASH diet, the low GI diet, or the Western-style diet. Testing will again be conducted after 2 weeks of weight stability on the study diet. Testing will include the assessment of insulin sensitivity and other metabolic parameters, such as blood sugar and cholesterol levels, blood pressure, and inflammation. This study will provide important information about the effects of these promising dietary patterns on features of the metabolic syndrome, in the absence of weight loss.

ELIGIBILITY:
Inclusion Criteria:

1. Nonsmoking men and postmenopausal women, ages 18 - 65. Premenopausal women who would not be expected to have significant fluctuations in estrogen and progesterone levels during the study (e.g. those on continuous monophasic hormonal contraception) may be included in the study at the discretion of the PI or designated study staff.
2. Body mass index (BMI) of at least 27 kg/m2
3. Body weight < 200 kg (the weight limit of the Bod Pod® scale)
4. Evidence of insulin resistance, as suggested by any one of the following:

   * Fasting glucose of 100 mg/dL or higher
   * Impaired glucose tolerance, with a glucose concentration of 140 mg/dL or higher, 2 hours after a 75-gram oral glucose challenge.
   * A fasting insulin concentration of 9 mIU/L or higher
5. Willingness to consume only study food and drink for the duration of the study
6. Willingness to be randomized to any one of the three study diets
7. If applicable, willingness to maintain consistent intake of coffee and/or tea during the inpatient periods (due to the potential effects of these drinks on inflammatory markers)
8. Willingness to avoid the use of all over-the-counter or prescription vitamins, dietary supplements, and herbal products during the study. At the PI's discretion, other nutritional supplements, such as iron, may also be continued during the study if they are deemed medically necessary and are unlikely to influence study results.
9. If applicable, willingness to continue current antihypertensive medications (especially angiotensin converting enzyme inhibitors and angiotensin receptor blockers, which may affect levels of inflammatory markers) at the same dose and schedule throughout the study,unless a change is advised by the subject's primary care provider or the study investigators
10. Willingness to avoid the use of non-steroidal anti-inflammatory drugs (NSAIDS), including low-dose daily aspirin, throughout the inpatient admission, (due to the potential effects of these agents on inflammatory markers).
11. at least two of the following:

    * waist circumference greater than 35" in women or 40" in men
    * blood pressure greater than 120/80 mmHg but less than 150/90 mmHg (on 2 blood pressure medications or less)
    * triglyceride level greater than 150 but less than 500 mg/dL
    * HDL ("good") cholesterol less than 40 mg/dL in men or 50 mg/dL in women

Exclusion Criteria:

1. Current tobacco smoking
2. History of a bleeding disorder
3. Known or suspected cardiovascular disease, including angina, myocardial infarction, medical or surgical treatment for atherosclerotic disease, arrhythmia, or congestive heart failure
4. Blood pressure higher than 145/90 after 10 minutes of rest, confirmed on two or more visits, or treatment with three or more antihypertensive agents at any blood pressure. Subjects taking up to two antihypertensive agents may be included in the study if 1) BP is at least 115/75 mmHg but < 145/90 mmHg on these agents and 2) they agree to remain on the same medications (and same dosages) during the study, unless otherwise advised by a primary care provider or study investigators (e.g. the dosage may be reduced or the medication may be stopped if signs or symptoms of hypotension develop during the study)
5. Fasting glucose > 165 mg/dL, glycosylated hemoglobin > 8%, or any treatment with oral hypoglycemic agents, insulin sensitizing agents (e.g. metformin or thiazolidinediones), insulin, incretin mimetics (e.g. exenatide), amylin analogues (e.g. pramlintide), or endocannabinoid receptor antagonists (e.g. rimonabant). Volunteers with type 2 diabetes and a glycosylated hemoglobin level of 7.5% or higher will be encouraged to discuss treatment options (e.g. pharmacotherapy versus study participation) with their primary care providers before enrolling in the study
6. History of chronic glucocorticoid use, oral glucocorticoid use for more than 5 days in the previous year, or anticipated treatment with oral or intravenous glucocorticoids during the study period. Daily, low-dose, inhaled or nasal glucocorticoids may be acceptable in some cases, at the discretion of the Principal Investigator.
7. Current treatment with over-the-counter or prescription weight loss medications, such as orlistat or sibutramine
8. History of bariatric surgery
9. Current treatment with any cholesterol-lowering medications, such as statins, niacin,fibrates, or ezetimibe
10. Hyperthyroidism or untreated hypothyroidism. Subjects with chronic, treated, stable hypothyroidism may be included in the study at the discretion of the Principal Investigator
11. Obstructive sleep apnea, or significant symptoms suggestive of this condition
12. Active gallstone disease
13. Known history of chronic hepatitis, or liver enzymes (AST or ALT) more than 2.5 times the upper limit of normal
14. Known infection with HIV or confirmed positive test for HIV antibody
15. Inflammatory bowel disease, active cancer, or any other medical condition that may cause significant acute weight loss or gain
16. Sustained weight loss > 5% of body weight in the previous two months, or sustained weight loss > 10% of body weight in the previous six months
17. History of kidney stones
18. Chronic or acute renal disease
19. Serum calcium, potassium, or magnesium above the normal limit, confirmed on two screening tests
20. Seizure disorder
21. History of any inpatient psychiatric admission within the past two years
22. History of schizophrenia, psychosis, or bipolar disorder
23. History of anorexia nervosa or bulimia nervosa, as defined in the Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV), or a history of medical or psychological treatment for an eating disorder
24. Severe binge eating disorder, as defined as a Binge Eating Scale score of 27 or more. Individuals with scores of 18-26, which may be indicative of moderate eating disturbances, will be evaluated further to determine whether moderate to severe eating pathology actually exists. This evaluation process will be based on the DSMIVresearch criteria for binge eating disorder. Individuals with scores of 18-26 who meet the DSM-IV research criteria for binge eating disorder will be excluded, whereas those without significant eating pathology may be included in the study.
25. Untreated moderate to severe depression, as evidenced by a Beck Depression Inventory score of 20 or higher at screening. Subjects with a remote history of depression or stable, treated depression may be included in the study at the discretion of the Principal Investigator
26. History of alcohol or drug abuse within the previous two years
27. History, physical, or laboratory findings suggestive of any other medical or psychological condition that would, in the opinion of the principal investigator, make the candidate ineligible for the study.
28. Any social or behavioral condition that, in the opinion of the investigator, would interfere with adherence to study requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in hepatic insulin sensitivity from the first testing battery (on Western diet) to the second testing battery (on study diet). Hepatic insulin sensitivity will be assessed using the homeostatic model assessment plasma | 3 years

SECONDARY OUTCOMES:
Peripheral (muscle) insulin sensitivity, Glycemic control,Glycemic responses to a representative breakfast, Systemic inflammation, blood endotoxin levels, lipids, Systolic and diastolic blood pressure, body composition, and dietary satisfaction. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Neff, MD, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States